CLINICAL TRIAL: NCT02407600
Title: Phase II, Double-blind, Placebo-controlled, Crossover Study Evaluating a 5HT3 Antagonist Plus Dexamethasone With or Without Fosaprepitant in Patients With Advanced NSCLC Receiving Carboplatin Based Chemotherapy
Brief Title: Study Assessing Fosaprepitant in Advanced NSCLC Patients Treated With Carboplatin Based Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ajeet Gajra (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Ajeet Gajra, Associate Professor, State University of New York - Upstate Medical University
Organization: State University of New York - Upstate Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Merck-50437
Record Dates: First submitted 2015-03-20; First posted 2015-04-03 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Non-small Cell Lung Cancer; Vomiting; Nausea; Emesis
Keywords: EMEND for Injection; 5HT-3; Fosaprepitant
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Vomiting; Nausea | interventions — fosaprepitant; Aprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fosparepitant administered in 1st cycle (Active Comparator): Fosaprepitant (Emend) for Injection 150 mg is administered, one time, intravenously on day 1 only, as an infusion with a duration of 30 minutes. It will be initiated approximately 30 minutes prior to the subjects first chemotherapy cycle. An intravenous saline placebo will be administered on day 1 of the second chemotherapy cycle, in the same manor as EMEND for Injection.
  Interventions: Drug: FOSAPREPITANT (Emend); Drug: Placebo
- Fosaprepitant administered in 2nd cycle (Sham Comparator): Subject will receive a saline Placebo intravenously on day 1 of their first chemotherapy cycle. For the subject's second chemotherapy cycle, EMEND for Injection 150 mg is administered, one time, intravenously on day 1, as an infusion with a duration of 30 minutes. It will be initiated approximately 30 minutes prior to the subjects second chemotherapy cycle.
  Interventions: Drug: FOSAPREPITANT (Emend); Drug: Placebo

INTERVENTIONS:
Drug: FOSAPREPITANT (Emend) — Uee of fosprepitant in EITHER first OR 2nd cycle of carboplatin containing combination chemotherapy in patients with advanced NSCLC
  Other Names: EMEND for Injection
Drug: Placebo

SUMMARY:
This study evaluates the addition of fosaprepitant to currently available antiemtic treatments of carboplatin chemotherapy-induced nausea and vomiting in advanced non-small cell lung cancer patients. Half of the patients will receive fosaprepitant in their first chemotherapy cycle, and a placebo on their second chemotherapy cycle. The other half of the patients will begin their first chemotherapy cycle.

DETAILED DESCRIPTION:
The addition of aprepitant to 5HT-3 antagonist and steroid is approved for the prevention of acute and delayed nausea for highly emetogenic chemotherapy (HEC). The use of oral aprepitant 3 day regimen has been evaluated in moderately emetogenic chemotherapy. However, its use has not been explored in carboplatin containing combination regimens in advanced non-small cell lung cancer (NSCLC). An equivalency study compared fosaprepitant, a 1-day intravenous formulation of aprepitant, with oral aprepitant. Findings demonstrate equivalence between the agents for complete response and both emesis and nausea control. Fosaprepitant was endorsed by the ASCO Update Committee as an acceptable NK1 receptor antagonist. However, there has been no evaluation of this iv formulation with moderately emetogenic chemotherapy and specifically carboplatin containing regimens in NSCLC. Therefore, the investigators propose a double-blind, randomized placebo controlled cross-over phase II study assessing the role of fosaprepitant in the prevention of nausea and emesis in patients receiving carboplatin based chemotherapy for advanced NSCLC.

Patients will be treated with Emend/ placebo administered intravenously on day 1 of cycles 1 of carboplatin based chemotherapy with crossover to the alternate agent (placebo/ Emend) on day 1 of cycle 2 with each cycle being 21 days. Fosaprepitant will be administered intravenously on day 1 of either cycle 1 or cycle 2 prior to carboplatin based chemotherapy. Placebo will be administered as the alternative agent. Study team and the subject will be blinded to fosaprepitant versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patient age > 18 years and able to sign informed consent.
* ECOG PS 0-2
* Patients with stage IV or recurrent NSCLC being treated with carboplatin based regimen with palliative intent.
* Acceptable chemotherapy regimens include:
* Carboplatin (AUC of 5 OR 6) q 21 days with:

  * Paclitaxel Q 21 days OR
  * Docetaxel Q 21 days OR
  * Pemetrexed Q 21 days (non-squamous histology with Vitamin B12 and folate supplementation) OR
  * Gemcitabine administered days 1 and 8 Q 21 days OR
  * Vinorelbine administered days 1 and 8 Q 21 days
* The addition of bevacizumab to chemotherapy is permitted where indicated and clinically appropriate.
* Patients who have received prior adjuvant chemotherapy for lung cancer ( > 1 year prior) and have recurred are eligible if it has been > 1 year since completion of adjuvant chemotherapy.
* Patients who have been treated for locally advanced lung cancer with concurrent chemoradiation but completed such therapy > 1 year ago are eligible provided they meet all other inclusion criteria.
* Patients who have received prior adjuvant chemotherapy for lung cancer ( > 1 year prior) and have recurred are eligible if it has been > 1 year since completion of adjuvant chemotherapy.
* Patients who have been treated for locally advanced lung cancer with concurrent chemoradiation but completed such therapy > 1 year ago are eligible provided they meet all other inclusion criteria.
* Laboratory parameters:
* Serum creatinine < 2.0 and
* AST, ALT < 3 time the upper limit of normal
* Platelet count ≥ 100,00/cumm
* ANC ≥ 1500/ cumm on day of therapy (day # 1 of the cycle)
* Hemoglobin > 8.0 g/dl

Exclusion Criteria:

* History of allergic reaction to aprepitant or fosaprepitant
* Use of other investigational agents concurrently with chemotherapy
* Uncontrolled systemic hypertension with SBP > 180 and/ or DBP> 110
* Concurrent use of pimozide, terfenadine, astemizole, or cisapride (fosaprepitatnt is a dose-dependent inhibitor of cytochrome P450 isoenzyme 3A4 (CYP3A4). If used concurrently with above agents, there can be elevated plasma concentrations of these drugs, potentially causing serious or life-threatening reactions. Patients may be enrolled on the study if at least 7 days have elapsed since last dose of such a medication.
* Women who are pregnant or lactating are not eligible. Women of childbearing age musthave a negative pregnancy test within 3 days of treatment and agree to use of contraception during the study period.
* Use of any of the CYP450 inducers like phenytoin, carbamazepine, barbiturates, rifimapicin, rifabutin or St John's wort within 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Assess the impact of addition of fosaprepitant upon the complete response (C.R.) rate (no emetic episodes or use of rescue medications) in patients with advanced NSCLC receiving carboplatin-based combination chemotherapy. | Days 1-5 following the first two cycles of carboplatin based combination chemotherapy
  The primary end point of the study is to determine the proportion of patients in each of the two groups (placebo and fosaprepitant) who achieve a CR, defined as no vomiting, no retching and no rescue therapy during days 1-5 following the first two cycles of carboplatin based combination chemotherapy using an intent to-treat (ITT) analysis.

SECONDARY OUTCOMES:
No emesis (defined as no emetic episodes regardless of use of rescue therapy) | Collection of data at the completion of 2 cycles, day 42.
  No emesis (defined as no emetic episodes regardless of use of rescue therapy)
Asses nausea based on visual analog scale (VAS) | Collection of data at the completion of 2 cycles, day 42.
  Assessment of nausea based on visual analog scale (VAS) and symptoms measured by M. D. Anderson Symptom Inventory to capture the following end points:
  1. No nausea (maximum VAS <5 mm on a 0 to 100 mm scale)
  2. No significant nausea (maximum VAS <25 mm on a 0 to 100 mm scale)
  3. Complete protection (defined as no emetic episodes, no use of rescue therapy, and a maximum nausea visual analogue scale [VAS] score <25 mm on a 0 to 100 mm scale)
Patient's preferred cycle | Collection of data at the completion of 2 cycles, day 42.
  After the 2 cycles, determine patient's stated preferred cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Ajeet Gajra, MD FACP, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

REFERENCES:
- [Background] Fernandez-Ortega P, Caloto MT, Chirveches E, Marquilles R, Francisco JS, Quesada A, Suarez C, Zorrilla I, Gomez J, Zabaleta P, Nocea G, Llombart-Cussac A. Chemotherapy-induced nausea and vomiting in clinical practice: impact on patients' quality of life. Support Care Cancer. 2012 Dec;20(12):3141-8. doi: 10.1007/s00520-012-1448-1. Epub 2012 Mar 31. PMID 22460057
- [Background] Wheatley-Price P, Le Maitre A, Ding K, Leighl N, Hirsh V, Seymour L, Bezjak A, Shepherd FA; NCIC Clinical Trials Group. The influence of sex on efficacy, adverse events, quality of life, and delivery of treatment in National Cancer Institute of Canada Clinical Trials Group non-small cell lung cancer chemotherapy trials. J Thorac Oncol. 2010 May;5(5):640-8. doi: 10.1097/JTO.0b013e3181d40a1b. PMID 20354457
- [Background] Hesketh PJ, Kris MG, Grunberg SM, Beck T, Hainsworth JD, Harker G, Aapro MS, Gandara D, Lindley CM. Proposal for classifying the acute emetogenicity of cancer chemotherapy. J Clin Oncol. 1997 Jan;15(1):103-9. doi: 10.1200/JCO.1997.15.1.103. PMID 8996130
- [Background] Grunberg SM, Warr D, Gralla RJ, Rapoport BL, Hesketh PJ, Jordan K, Espersen BT. Evaluation of new antiemetic agents and definition of antineoplastic agent emetogenicity--state of the art. Support Care Cancer. 2011 Mar;19 Suppl 1:S43-7. doi: 10.1007/s00520-010-1003-x. Epub 2010 Oct 24. PMID 20972805